CLINICAL TRIAL: NCT00075959
Title: CHANT (Cerebral Hemorrhage And NXY Treatment) A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multicenter, Phase IIb Study to Assess the Safety and Tolerability of Intravenous Infusion of NXY-059 in Adult Patients With Acute Intracerebral Hemorrhage (ICH)
Brief Title: Safety of NXY-059 for the Treatment of Patients Who Have Suffered From a Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: SA-NXY-0012; 0012; CHANT
Record Dates: First submitted 2004-01-12; First posted 2004-01-14 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: Stroke; cerebral vascular accident; CVA; Hemorrhage; Intracerebral Hemorrhage (ICH); Brain Attack; Cataplexy
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hemorrhage; Cataplexy | interventions — disufenton sodium

INTERVENTIONS:
Drug: NXY-059

SUMMARY:
This study will determine if NXY-059 is safe in patients with an acute stroke caused by bleeding in the central nervous system. The primary objective was to assess the safety and tolerability of NXY-059 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Intracerebral Hemorrhage as the cause of stroke symptoms
* Onset of symptoms within 6 hours
* Full functional independence prior to the present stroke

Exclusion Criteria:

* Unconsciousness
* Subjects who are unlikely to complete the infusion of investigational product and/or are unlikely to undergo active medical management during that period due to a severe clinical condition.
* Severe illness with life expectancy less than 6 months.
* Known severe kidney disorder.
* Current known alcohol or illicit drug abuse or dependence.
* Pregnant or breast-feeding.
* Treatment with acetazolamide and methotrexate is not permitted during the infusion
* Participation in a previous clinical study within 7 days.
* Meets all other exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Global disability on modified Rankin scale at 90 days

SECONDARY OUTCOMES:
NIH stroke scale
Barthel Index
Stroke Impact Scale

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca NXY-059 Medical Science Director, MD, Study Director — AstraZeneca
Locations (64):
- United States (64):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Carmichael, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Santa Rosa, California
  - Research Site, Walnut Creek, California
  - Research Site, Danbury, Connecticut
  - Research Site, Melbourne, Florida
  - Research Site, Ocala, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Punta Gorda, Florida
  - Research Site, Tampa, Florida
  - Research Site, Weston, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Duluth, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Arlington Heights, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Marrero, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, South Weymouth, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, East Lansing, Michigan
  - Research Site, Robbinsdale, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Reno, Nevada
  - Research Site, Edison, New Jersey
  - Research Site, Holmdel, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Ridgewood, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Manhasset, New York
  - Research Site, Schenectady, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Abington, Pennsylvania
  - Research Site, Danville, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Bristol, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Virginia Beach, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Marshfield, Wisconsin